CLINICAL TRIAL: NCT03806517
Title: Bone Mineral Density in Tremor Dominant Type Compared to Postural Instability Gait Difficulty Type Parkinson's Disease: a Cross-sectional Study
Brief Title: Bone Mineral Density Changes Among Clinical Subtypes of Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Head of Department of Physiotherapy and Rehabilitation, Ordu University
Other Study IDs: Ordu University 1
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease; Bone Loss
Keywords: bone mineral density; Parkinson's disease; tremor; postural instability and gait difficulty; akinetic-rigid
MeSH Terms: conditions — Parkinson Disease; Bone Diseases, Metabolic; Tremor; Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tremor dominant type group: Tremor dominant type (TDT) group will consist of the patients with tremor premotor symptoms.
- PIGD dominant type group: Postural instability and gait difficulty dominant type (PIGDT) group will consist of the patients with axial premotor symptoms.
- Healthy control group: Healthy control group will consist of the subjects with same age and sex matched individuals in PD group.

SUMMARY:
The bone loss in Parkinson's disease (PD) emerges as a non-motor symptom with motor and non-motor outcomes, such as fracture and musculoskeletal pain. Bone mineral density (BMD) is decreasing in patients with PD when compared to sex and age-matched healthy controls. The changes in BMD according to clinical subtypes of PD is unknown. The investigators are planning to compare the BMD status between the tremor dominant and postural instability and gait difficulty type of PD.

DETAILED DESCRIPTION:
The investigators are planning to complete this study between January and February 2019. This study will be performed at Ordu University Education and Research Hospital, Neurology Department.

All patients admitted to the outpatient clinic will be evaluated in terms of inclusion criteria. The control group consisted of people who do not have any orthopedic, neurological or metabolic disorders which may affect the BMD.

ELIGIBILITY:
For TDT and PIGDT PD group

Inclusion Criteria:

Clinical diagnosis of idiopathic Parkinson's disease Age of 40-85 years

Exclusion Criteria:

Having additional orthopedic and neurological disorders Having metabolic disease, Having steroid drug use

For Control group

The similar age and sex-matched healthy individuals who have no orthopedic, metabolic and neurological disorders, and steroid use will be included in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The PD group will be selcted from Neurology Department, Movement Disorders Clinic.
  The control group will be selected from community population.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-02-10 (Estimated); Primary Completion 2019-02-25 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry (DEXA) | 10-15 minutes
  Bone mineral density will be dertermined using DEXA results. The results will be interpreted by WHO (World Health Organization) criteria.
  : T-score (T-score) is determined by DEXA method. A T-score value of more than minus means that there is excess bone loss.
  * Obsolete osteoporosis: A T-score of less than -2.5 SD and a history of fracture in a patient.
  * Osteoporosis: T-score below -2.5 SD. (Like -3, -4 ...)
  * Osteopenia: T-score between -1 and -2.5 SD
  * Normal: T-score value better than -1

SECONDARY OUTCOMES:
Hoehn and Yahr Scale | 2 minutes
  Disease progression will be assessed with Hoehn and Yahr Scale. The original scale included stages 1 through 5.
  Stage 0: No signs of disease.
  Stage 1: Unilateral symptoms only.
  Stage 2: Bilateral symptoms. No impairment of balance.
  Stage 3: Balance impairment. Mild to moderate disease. Physically independent.
  Stage 4: Severe disability, but still able to walk or stand unassisted.
  Stage 5: Needing a wheelchair or bedridden unless assisted.
Unified Parkinson's Disease Rating Scale (UPDRS) - Section of Activities of Daily Living (ADL) | 10 minutes
  The UPDRS- ADL section evaluates the impact of Parkinson disease on ADL according to patient's perspective. The ADL section consists of 13 items for gathering information on the patient's own perception of functional impairment due to PD. Each item scores between 0-4. 0 means normal and 4 means severe impairment. The total score change between 0-52. High scores indicate severe impairment.
Unified Parkinson's Disease Rating Scale (UPDRS) - Motor Section | 10 minutes
  Motor section of UPDRS determines the impairment due to the Parkinson's disease. Rigidity, bradykinesia and tremor items which are relating with upper extremity function will be assessed. Each item scores between 0-4. 0 means normal and 4 means severe impairment. The total score change between 0-56.
Unified Parkinson's Disease Rating Scale (UPDRS) - non-motor Section | 5 minutes
  Non-motor section of UPDRS evaluates the impact of the non motor symptoms in PD. Each item scores between 0-4. 0 means normal and 4 means severe impairment. Total score changes between 0-52.
Unified Parkinson's Disease Rating Scale (UPDRS) - complications Section | 5 minutes
  Complications section of UPDRS evaluates the complications after the levodopa treatment in PD. Each item scores between 0-4. 0 means normal and 4 means severe impairment. Total score changes between 0-24.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim ACARÖZ CANDAN, Principal Investigator — Ordu University
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)